CLINICAL TRIAL: NCT05298189
Title: Understanding How Cognitive Performance and Physiological Measures Change After Acute Stress and How Different Sensory Features of a Relaxation Room Help Recover
Brief Title: Acute Stress Recovery
Acronym: ASR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Well Living Lab, Inc. (Industry)
Collaborators: Mayo Clinic (Other); Delos Living LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB 21-005885
Record Dates: First submitted 2022-03-03; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Audio-visual Group (Experimental)
  Interventions: Behavioral: MindBreaks - Audio-visual
- Auditory-only Group (Experimental): This group will recover in the relaxation room with only auditory stimuli.
  Interventions: Behavioral: MindBreaks - Auditory-only
- Visual-only group (Experimental)
  Interventions: Behavioral: MindBreaks - Visual-only
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: MindBreaks - Audio-visual — A "MindBreaks" room is designed to deliver short, effective, and restorative breaks to help increase energy, reduce stress, enhance mood, improve focus, and boost performance. For this intervention, the MindBreaks room will contain visual and auditory stimuli.
  Arms: Audio-visual Group
Behavioral: MindBreaks - Auditory-only — A "MindBreaks" room is designed to deliver short, effective, and restorative breaks to help increase energy, reduce stress, enhance mood, improve focus, and boost performance. For this intervention, the MindBreaks room will contain only auditory stimuli.
  Arms: Auditory-only Group
Behavioral: MindBreaks - Visual-only — A "MindBreaks" room is designed to deliver short, effective, and restorative breaks to help increase energy, reduce stress, enhance mood, improve focus, and boost performance. For this intervention, the MindBreaks room will contain only visual stimuli.
  Arms: Visual-only group

SUMMARY:
The proposed study aims to evaluate whether different features of a relaxation room affect how individuals recover from acute stress. This study will use a unique methodology to capture participants' physiological and behavioral measures through a combination of non-invasive technologies, including wearables devices, active sensors, cognitive tasks, and/or subjective questionnaires. Participants will perform a stress induction task, after which they will rest in a relaxation room. Physiological measures and cognitive performance will be recorded throughout the experiment to determine whether features of the relaxation room promote recovery after acute stress. Identifying the occurrence of stress and ways to potentially reduce the effects of stress could lead to novel interventions for helping individuals reduce work-related stress.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least age 18
2. Participants are able to remain in the Well Living Lab for 3-4 hours
3. Participants are able to perform scripted tasks
4. Participants are able to provide informed consent
5. Participants are able to wear the wearable devices at all times during the study
6. Participants have completed a COVID vaccine regimen and can provide written documentation verifying vaccination status at least fourteen (14) days prior to the commencement of the research study

Exclusion Criteria:

1. Participants with a reported history of diagnosed mood, anxiety, or major health disorders
2. Participants who have used steroid-based medications within the past three years
3. Participants with a history of drug/alcohol abuse
4. Participants with or recovering from nicotine dependency who cannot use a nicotine patch
5. Participants who consume excessive amounts of caffeine
6. Participants who have had severe sleep disturbance (e.g., shift work, chronic insomnia)
7. Women who are pregnant or intend to become pregnant at the time of the study
8. Participants with a history of diagnosed cognitive impairment
9. Participants taking any medications that might affect the physiological measures of interest
10. Participants with anything that might affect collecting the physiological measures of interest (e.g., cosmetic products, head coverings, head products, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive performance relative to baseline | throughout the one day experimental session at time points approximately -35 minutes, -5 minutes, +15 minutes, +35 minutes, +55 minutes relative to the start of the stress induction task
  Participants will perform the operational SPAN (OSPAN) and symmetry SPAN (SSPAN) working memory assessments at 5 time points throughout the experimental session. The unit score and load score from these assessments are used to measure changes in working memory cognitive performance. Measurements are taken at approximately -35 minutes, -5 minutes, +15 minutes, +35 minutes, and +55 minutes relative to the start of the stress induction task (Trier social stress test, TSST). Each measure will be compared with the -35 minute baseline measurement to detect a change in performance.
  [Note: times are approximate as there might be slight temporal changes due to the self-paced duration it takes each participant to complete certain portions of the experiment].
Change in perceived stress relative to baseline | throughout the one day experimental session at time points approximately -35 minutes, -5 minutes, +5 minutes, +15 minutes, +35 minutes, +55 minutes relative to the start of the stress induction task
  Measures of perceived stress from self-reported surveys will be compared before, during and after a stress induction task relative to baseline. Surveys are completed after the cognitive assessments and during the stress induction task. Measurements are taken at approximately -35 minutes, -5 minutes, +5 minutes, +10 minutes, +15 minutes, +35 minutes, and +55 minutes relative to the start of the stress induction task (Trier social stress test, TSST). Each measure will be compared with the -35 minute baseline measurement to detect a change in performance.
  [Note: times are approximate as there might be slight temporal changes due to the self-paced duration it takes each participant to complete certain portions of the experiment].
Change in heart rate relative to baseline | throughout the one day experimental session during baseline (-35 minutes to -5 minutes), stress induction task (+0 to +15 minutes), recovery period #1 (+15 to +35 minutes), recovery period #2 (+35 to +55 minutes) epochs
  Measures of heart rate from wearable devices will be compared before, during and after a stress induction task. Heart rate will be measured continuously and binned during the following epochs of the experimental session (all times relative to the start of the stress induction task and are approximates due to some temporal delays in transitioning between epochs): baseline (-35 minutes to -5 minutes), stress induction task (+0 to +15 minutes), recovery period #1 (+15 to +35 minutes), recovery period #2 (+35 to +55 minutes).
  [Note: times are approximate as there might be slight temporal changes due to the self-paced duration it takes each participant to complete certain portions of the experiment].
Change in electroencephalography (EEG) alpha band power relative to baseline | throughout the one day experimental session during baseline (-35 minutes to -5 minutes), stress induction task (+0 to +15 minutes), recovery period #1 (+15 to +35 minutes), recovery period #2 (+35 to +55 minutes) epochs
  Measures of neural activity, (electroencephalography, EEG) from a wearable device will be compared before, during and after a stress induction task. Alpha band power will be measured and binned during the following epochs of the experimental session (all times relative to the start of the stress induction task and are approximates due to some temporal delays in transitioning between epochs): baseline (-35 minutes to -5 minutes), stress induction task (+0 to +15 minutes), recovery period #1 (+15 to +35 minutes), recovery period #2 (+35 to +55 minutes).
  [Note: times are approximate as there might be slight temporal changes due to the self-paced duration it takes each participant to complete certain portions of the experiment].

CONTACTS AND LOCATIONS:
Locations (1):
- Well Living Lab Inc., Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No